CLINICAL TRIAL: NCT04308590
Title: Glucocorticoid Receptor Antagonism in the Treatment of Hypercortisolism in Patients With Cortisol-Secreting Adrenal Adenomas or Hyperplasia (GRADIENT): A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Relacorilant
Brief Title: A Study of the Efficacy and Safety of Relacorilant in Patients With Cortisol-Secreting Adrenal Adenomas
Acronym: GRADIENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT125134-456
Record Dates: First submitted 2020-02-27; First posted 2020-03-16 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypercortisolism
Keywords: Cushing syndrome; Cushing; Hypercortisolemia; Type 2 Diabetes; Impaired Glucose Intolerance; Hypertension; Adrenocorticotropic hormone; Primary Pigmented Nodular Adrenal Disease; Macronodular adrenal hyperplasia; Adrenal Adenoma; Adrenal Autonomy; Cortisol; Autonomous cortisol secretion
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic; Diabetes Mellitus, Type 2; Hypertension | interventions — relacorilant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Relacorilant (Experimental): Patients will receive relacorilant increased sequentially from 100 mg once daily to a maximum dose of 400 mg once daily.
  Interventions: Drug: Relacorilant; Other: Placebo
- Placebo (Placebo Comparator): Patients will receive placebo matched to study drug once daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Relacorilant — Relacorilant is supplied as blister-packed capsules for oral dosing. Relacorilant 400 mg dose consists of 4 relacorilant 100-mg capsules. Relacorilant 100-mg, 200-mg, and 300-mg doses are each given as a combination of 4 capsules containing relacorilant 100-mg and placebo as per the assigned dose.
  Other Names: CORT125134
  Arms: Relacorilant
Other: Placebo — Placebo is supplied as blister-packed capsules for oral dosing. Each dose consists of 4 capsules containing placebo.

SUMMARY:
This is a Phase 3, randomized, double-blind, placebo-controlled study to assess the efficacy, and safety of relacorilant to treat hypercortisolism in patients with cortisol-secreting adrenal adenoma or hyperplasia associated with diabetes mellitus/ impaired glucose tolerance (DM/IGT) and/or uncontrolled systolic hypertension (HTN).

DETAILED DESCRIPTION:
The primary outcome measures of the study are 1) to assess the efficacy of relacorilant based on blood pressure control at Week 22 compared with placebo, and 2) to assess the safety of relacorilant based on adverse events. Patients will be randomized in a 1:1 ratio to treatment with relacorilant (active drug) or placebo. Patients will receive relacorilant or placebo for 22 weeks. Patients who complete the study may also be eligible to roll over into an extension study.

ELIGIBILITY:
Inclusion Criteria:

* Shows lack of cortisol suppression on dexamethasone suppression test
* Suppressed or low early-morning adrenocorticotropic hormone (ACTH) levels
* A radiologically confirmed adrenal lesion
* Has IGT or DM
* Has uncontrolled HTN

Exclusion Criteria:

* Has severe, uncontrolled HTN
* Has poorly controlled DM
* Has DM Type 1
* Has significantly abnormal liver test results or severe renal insufficiency
* Has uncontrolled, clinically significant hypothyroidism or hyperthyroidism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Moraitis, MD, Study Director — Corcept Therapeutics
Locations (45):
- United States (22):
  - Site 27, Birmingham, Alabama
  - Site 17, Stanford, California
  - Site 53, Torrance, California
  - Site 07, Atlanta, Georgia
  - Site 16, Indianapolis, Indiana
  - Site 09, Metairie, Louisiana
  - Site 36, Baltimore, Maryland
  - Site 11, Fall River, Massachusetts
  - Site 33, Rochester, Minnesota
  - Site 06, Jackson, Mississippi
  - Site 54, Reno, Nevada
  - Site 10, Jamaica, New York
  - Site 44, New York, New York
  - Site 01, Wilmington, North Carolina
  - Site 30, Cleveland, Ohio
  - Site 21, Columbus, Ohio
  - Site 02, Summerville, South Carolina
  - Site 20, Dallas, Texas
  - Site 03, El Paso, Texas
  - Site 05, Fort Worth, Texas
  - Site 08, Houston, Texas
  - Site 15, Spokane, Washington
- Site 25, Vienna, Vienna, Austria
- Site 22, Sofia, Bulgaria
- Germany (2):
  - Site 50, Munich, Bavaria
  - Site 46, Würzburg
- Israel (2):
  - Site 32, Ramat Gan
  - Site 23, Tel Aviv
- Italy (8):
  - Site 40, Milan, Milano
  - Site 31, Rome, Roma
  - Site 43, Orbassano, Torino
  - Site 34, Milan
  - Site 28, Napoli
  - Site 51, Padua
  - Site 37, Rome
  - Site 52, Torino
- Poland (3):
  - Site 48, Gliwice
  - Site 47, Krakow
  - Site 35, Lublin
- Romania (3):
  - Site 42, Bucharest
  - Site 38, Bucharest
  - Site 41, Bucharest
- Spain (3):
  - Site 14, Málaga
  - Site 13, Seville
  - Site 26, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 307 patients were screened and 137 were enrolled.
Period: Overall Study
Arm/Group | Relacorilant | Placebo
Started | 68 | 69
Completed | 43 | 61
Not Completed | 25 | 8
Not completed — Adverse Event | 12 | 2
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Subject does not want to continue with Pi | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was patients in the Intent-to-treat (ITT) Population which included all randomized patients, even if they did not receive any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relacorilant | Placebo | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.11) | 63.0 (9.00) | 62.7 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 64 | 63 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 63 | 65 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Hypertension (HTN) only [Count of Participants; unit: Participants] — HTN without diabetes mellitus (DM) or impaired glucose intolerance (IGT). HTN is defined as average systolic blood pressure (SBP) ≥130 to ≤170 mm Hg based on 24-hour ambulatory blood pressure monitoring (ABPM).
  Participants | 20 | 21 | 41
Diabetes mellitus (DM) or impaired glucose tolerance (IGT) only [Count of Participants; unit: Participants] — DM/IGT without HTN. DM is defined as fasting plasma glucose ≥126 mg/dL and/or 2-hour oral glucose tolerance test (oGTT) plasma glucose ≥200 mg/dL, or hemoglobin A1C (HbA1c) ≥6.5%. IGT is defined as plasma glucose ≥140 mg/dL and <200 mg/dL at 2 hours on the 2-hour oGTT.
  Participants | 26 | 27 | 53
HTN and DM/IGT [Count of Participants; unit: Participants] — HTN and DM/IGT defined as above.
  Participants | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Change in Average 24-hour SBP
Description: Blood pressure was measured by 24-hour ABPM. The 24-hour average SBP is reported.
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had HTN with or without DM/IGT at Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 42 | 42
mm Hg | -5.56 [-10.459 to -0.659] | -2.89 [-6.794 to 1.006]
Statistical Analysis 1: Comparison: Relacorilant vs Placebo; Test type: Equivalence — The primary analysis will determine whether there is a difference between treatment groups in terms of change from Baseline to Week 22 in 24-hour average SBP. This was performed using a linear mixed-model-for-repeated-measures (MMRM) analysis using a placebo wash-out multiple imputation for treatment discontinuation and for patients that use rescue medication; p = 0.4160, Mixed Models Analysis; Least squares mean difference = -2.67, 95% CI 2-sided [-9.096 to 3.766]

2. Primary Outcome: Number of Patients With 1 or More Treatment-emergent Adverse Events (TEAEs) as Graded by CTCAE v5.0.
Time Frame: Baseline and up to Week 26
Population: The analysis population was patients in the Safety Population which included all randomized patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 68 | 69
Participants | 67 | 60

3. Secondary Outcome: Change in Area Under the Concentration-time Curve of Blood Glucose (AUCglucose)
Description: AUCglucose was calculated based on results of the plasma 2-hour oGTT.
Time Frame: Before and at time intervals up to 2 hours post glucose drink at Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had DM/IGT with or without HTN at Baseline and had an available assessment at Week 22.
Measure: Least Squares Mean (95% Confidence Interval); unit: hours x mmol/L
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 29 | 38
hours x mmol/L | -1.566 [-3.472 to 0.340] | 1.008 [-0.661 to 2.676]

4. Secondary Outcome: Change in Average Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured by 24-hour ABPM. Daytime average DBP was measured from 06:00 to 21:59. Nighttime average DBP was measure from 22:00 to 05:59.
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had HTN with or without DM/IGT at Baseline and had an available assessment at Week 22.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 21 | 30
mm Hg
  24-hour Average | -3.3 [-6.1 to -0.5] | -1.4 [-3.8 to 0.9]
  Daytime Average | -3.1 [-6.0 to -0.1] | -1.0 [-3.5 to 1.6]
  Nighttime Average | -3.0 [-6.4 to 0.5] | -0.6 [-3.5 to 2.4]

5. Secondary Outcome: Change in Average Heart Rate (HR)
Description: Heart rate was measured by 24-hour ABPM. Daytime average HR was measured from 06:00 to 21:59. Nighttime average HR was measure from 22:00 to 05:59.
Time Frame: Baseline and Week 22
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 21 | 30
Beats per minute
  24-hour Average | 2.0 [-0.4 to 4.5] | -2.0 [-4.1 to 0.1]
  Daytime Average | 1.7 [-1.1 to 4.5] | -1.5 [-3.9 to 0.9]
  Nighttime Average | 2.2 [-0.4 to 4.7] | -2.7 [-4.9 to -0.5]

6. Secondary Outcome: Change in Average Daytime and Nighttime SBP
Description: Blood pressure was measured by 24-hour ABPM. Daytime average SBP was measured from 06:00 to 21:59. Nighttime average SBP was measure from 22:00 to 05:59.
Time Frame: Baseline and Week 22
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 21 | 30
mm Hg
  Daytime Average | -4.5 [-9.0 to -0.1] | -2.5 [-6.3 to 1.4]
  Nighttime Average | -4.6 [-9.9 to 0.6] | -3.0 [-7.5 to 1.4]

7. Secondary Outcome: Change in Hemoglobin HbA1c for Patients With HbA1c ≥5.7% at Baseline
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had DM/IGT with HbA1c ≥5.7% at Baseline and had an available assessment at Week 22.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 25 | 36
Percentage | -0.29 [-0.49 to -0.09] | 0.00 [-0.17 to 0.17]

8. Secondary Outcome: Change in HbA1c for Patients With HbA1c ≥6.5% at Baseline
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had DM/IGT with HbA1c ≥6.5% at Baseline and had an available assessment at Week 22.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 11 | 17
Percentage | -0.57 [-1.00 to -0.14] | -0.19 [-0.52 to 0.14]

9. Secondary Outcome: Number of Patients With DM Who Achieved 2-hour oGTT Glucose <140 mg/dL
Description: Glucose was measured using the 2 hour timepoint of the 2-hour oGTT.
Time Frame: 2 hours post glucose drink at Week 22
Population: The analysis population was patients in the ITT Population who had DM with or without HTN at Baseline and had an available assessment at Week 22.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 27 | 28
Participants | 1 | 0

10. Secondary Outcome: Number of Patients With IGT Who Achieved 2-hour oGTT Glucose <140 mg/dL
Description: Glucose was measured using the 2 hour timepoint of the 2-hour oGTT.
Time Frame: 2 hours post glucose drink at Week 22
Population: The analysis population was patients in the ITT Population who had IGT with or without HTN at Baseline and had an available assessment at Week 22.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 18 | 16
Participants | 6 | 7

11. Secondary Outcome: Number of Patients With Any Dose Decrease in Antihypertensive Medication
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had HTN with or without DM/IGT at Baseline, received antihypertension medication both at Baseline and postbaseline, and had an available assessment at Week 22.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 22 | 33
Participants | 7 | 5

12. Secondary Outcome: Number of Patients With Any Dose Decrease in Diabetes Medication
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had DM/IGT at Baseline, received diabetes medication both at Baseline and postbaseline, and had an available assessment at Week 22.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 15 | 25
Participants | 0 | 0

13. Secondary Outcome: Number of Patients With Any Dose Increase or Switch in Antihypertensive Medication
Time Frame: Baseline and Week 22
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 22 | 33
Participants | 1 | 5

14. Secondary Outcome: Number of Patients With Any Dose Increase or Switch in Diabetes Medication
Time Frame: Baseline and Week 22
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 15 | 25
Participants | 4 | 3

15. Secondary Outcome: Number of Patients With HbA1c ≥6.5% at Baseline Who Achieved HbA1c <6.5%
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had DM with HbA1c ≥6.5% at Baseline and had an available assessment at Week 22.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 18 | 21
Participants | 3 | 4

16. Secondary Outcome: Number of Patients With Normalization of the 24-hour Average SBP (<130 mm Hg)
Description: Blood pressure was measured by 24-hour ABPM Test. Reported is the number of patients with HTN at Baseline who achieved SBP <130 mm Hg at Week 22.
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had HTN with or without DM/IGT at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 42 | 42
Participants | 9 | 13

17. Secondary Outcome: Number of Patients With a Reduction in 24-hour Average SBP by ≥5 mm Hg
Description: Blood pressure was measured by 24-hour ABPM. Reported is the number of patients with HTN at Baseline who achieved at least a 5 mm Hg reduction in 24-hour average SBP at Week 22.
Time Frame: Baseline and Week 22
Population: The analysis population was patients in the ITT Population who had HTN with or without DM/IGT at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant | Placebo
Number analyzed (Participants) | 42 | 42
Participants | 10 | 13

ADVERSE EVENTS:
Time Frame: Up to Week 26
Arm/Group | Relacorilant | Placebo
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/69
Serious Adverse Events (participants affected / at risk) | 15/68 | 4/69
Other Adverse Events (participants affected / at risk) | 65/68 | 60/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant (N=68) | Placebo (N=69)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant (N=68) | Placebo (N=69)
Abdominal pain upper (Gastrointestinal disorders) | 14 | 3
Nausea (Gastrointestinal disorders) | 13 | 8
Abdominal pain (Gastrointestinal disorders) | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Vomiting (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Fatigue (General disorders) | 16 | 10
Asthenia (General disorders) | 8 | 6
Oedema peripheral (General disorders) | 6 | 5
Dizziness (Nervous system disorders) | 10 | 4
Headache (Nervous system disorders) | 7 | 12
Sciatica (Nervous system disorders) | 5 | 1
Hypoaesthesia (Nervous system disorders) | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
COVID-19 (Infections and infestations) | 4 | 9
Urinary tract infection (Infections and infestations) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Hypertension (Vascular disorders) | 3 | 9
Insomnia (Psychiatric disorders) | 6 | 4
Anxiety (Psychiatric disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results, except as agreed with Corcept. The Investigator agrees to submit all manuscripts or abstracts to Corcept for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04308590/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04308590/SAP_001.pdf